CLINICAL TRIAL: NCT01971593
Title: Eplerenone to Prevent Myocardial Fibrosis in Congenital Heart Disease
Brief Title: The Effects of Eplerenone on Markers of Myocardial Fibrosis in Adult Congenital Heart Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Ari Cedars, Assistant Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WI170964
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Tetralogy of Fallot; Transposition of the Great Vessels With an Arterial Switch; Single Ventricle With a Fontan Palliation
MeSH Terms: conditions — Tetralogy of Fallot | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone after drug free period (Other): Patients will be given eplerenone 50mg for 12 months after an initial 3 month drug free period
  Interventions: Drug: Eplerenone
- Eplerenone before drug free period (Other): Patients will be given eplerenone 50mg for 12 months, followed by a 3 month drug free period
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone
  Other Names: Inspra

SUMMARY:
Hypothesis:

By blocking aldosterone signaling in patients with Tetralogy of Fallot, Transposition of the great vessels with a prior atrial switch, and single ventricle "Fontan" patients, incident heart failure will be delayed, symptoms of heart failure ameliorated, and risk of arrhythmias decreased through decreases in myocardial fibrosis.

Half of enrolled patients will complete an SF-36 quality of life questionnaire, perform a 6 minute walk, and have blood drawn for biomarker analysis at enrollment, again after 3 months without therapy, after 6 months on therapy, then finally after 12 months of eplerenone therapy. Half of enrolled patients will have the 3 month drug free period at the end of 12 months on therapy. Patients will be randomly assigned to drug free period up front versus at the conclusion of the trial period. Eplerenone will be started at a dose of 25mg and titrated up to 50mg at 4 weeks if tolerated. Blood will be drawn for basic metabolic panel analysis at enrollment, 3 months, 4 months to allow for dose titration, and at 6 and 12 months for monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of tetralogy of Fallot, transposition of the great vessels with a systemic right ventricle, or Fontan type palliation
* Patient followed regularly at Washington University-affiliated institution
* If female, willing to use 2 forms of contraception including one barrier method during protocol

Exclusion Criteria:

* GFR <30 ml/min
* Potassium >5.0 mmol/L
* Unable or unwilling to comply with study protocol
* Use of potassium sparing diuretics
* Use of an aldosterone blocker currently or previously
* Known intolerance of eplerenone or aldosterone blockade
* Pregnant, breastfeeding, or actively trying to get pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Eplerenone After Drug Free Period: Patients will be given eplerenone 50mg for 12 months after an initial 3 month drug free period
  Eplerenone
- Eplerenone Before Drug Free Period: Patients will be given eplerenone 50mg for 12 months, followed by a 3 month drug free period
  Eplerenone
Period: Overall Study
Arm/Group | Eplerenone After Drug Free Period | Eplerenone Before Drug Free Period
Started | 14 | 12
Completed | 9 | 8
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total Study Group: Crossover study, all patients pooled for baseline analysis
Arm/Group | Total Study Group
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17
Tetralogy of Fallot [Count of Participants; unit: Participants] | 12
Patients with Transposition of the Great Vessels with a Systemic Right Ventricle (RV) [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Procollagen N-terminal Peptide 1
Time Frame: Baseline, 6 months and 12 months from eplerenone administration
Population: Outcome analyzed only during the eplerenone period as specified in the protocol
Measure: Mean (Standard Deviation); unit: ug/ml
Groups:
- Total Study Group: Change from baseline at time of drug initiation
Arm/Group | Total Study Group
Number analyzed (Participants) | 17
ug/ml
  Baseline | 45.1 (15.4)
  6 Months | 48.9 (20.3)
  12 Months | 42.7 (12.2)

2. Primary Outcome: Procollagen III N-Terminal Peptide
Time Frame: Baseline, 6 months and 12 months from eplerenone administration
Population: Outcome analyzed only during the eplerenone period as specified in the protocol
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Total Study Group
Number analyzed (Participants) | 17
ug/ml
  Baseline | 4.6 (1.7)
  6 Months | 4.4 (1.5)
  12 Months | 4.4 (1.5)

3. Primary Outcome: Galectin 3
Time Frame: Baseline, 6 months and 12 months from eplerenone administration
Population: Outcome analyzed only during the eplerenone period as specified in the protocol
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Total Study Group
Number analyzed (Participants) | 17
ng/ml
  Baseline | 10.0 (2.4)
  6 Months | 11.6 (2.9)
  12 Months | 11.2 (2.2)

4. Secondary Outcome: 6 Minute Walk
Time Frame: Baseline, 6 months, 12 months from eplerenone administration
Population: Outcome analyzed only during the eplerenone period as specified in the protocol
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Total Study Group
Number analyzed (Participants) | 17
Feet
  Baseline | 1629 (261)
  6 Months | 1630 (250)
  12 Months | 1680.2 (255)

5. Secondary Outcome: Quality of Life
Description: Rand 36-item Short Score Physical Domain Scale (SF-36) Range: 0-100, Higher scores suggest better function
Time Frame: Baseline, 6 months, 12 months from eplerenone administration
Population: Outcome analyzed only during the eplerenone period as specified in the protocol
Measure: Mean (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Total Study Group
Number analyzed (Participants) | 17
Score on a scale
  Baseline | 87.5 [70 to 95]
  6 Months | 90 [75 to 97.5]
  12 Months | 85 [75 to 95]

6. Other Pre Specified Outcome: Serum Creatinine
Time Frame: Baseline, 6 months, 12 months from eplerenone administration
Population: Outcome analyzed only during the eplerenone period as specified in the protocol
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Total Study Group
Number analyzed (Participants) | 17
mg/dl
  Baseline | 0.9 (0.2)
  6 Months | 0.9 (0.2)
  12 Months | 0.9 (0.2)

ADVERSE EVENTS:
Time Frame: During 12 months while on eplerenone
Description: Adverse event data only collected during the eplerenone period
Groups:
- Eplerenone Period: Change from baseline at time of drug initiation
Arm/Group | Eplerenone Period
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 6/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eplerenone Period (N=26)
Leg cramping (Musculoskeletal and connective tissue disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)
hyperkalemia (Renal and urinary disorders) | 1 (1)
edema (Skin and subcutaneous tissue disorders) | 2 (2)
chest pain (Cardiac disorders) | 1 (1)
hypotension (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Incomplete study enrollment led to inadequate power to derive reliable conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No